CLINICAL TRIAL: NCT06950047
Title: Application of PediLoc®Locking Cannulated Blade Plate System in Distal Femoral Osteotomies - A Retrospective, Comparative Analysis of Consolidation Rates and Description of the Surgical Technique
Brief Title: PediLoc® Blade Plate in Distal Femoral Osteotomies
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Samuel Tschudi, Principal Investigator, University Children's Hospital, Zurich
Other Study IDs: 2025-0000
Record Dates: First submitted 2025-04-14; First posted 2025-04-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Osteotomy of Lower Extremity
Keywords: locking plate system; blade plate; distal femoral osteotomy; flexion contracture; deformities; multidimensional osteotomies; pediatric orthopedics; surgical technique
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- distal femoral osteotomies using the PediLoc® Locking Cannulated Blade Plate System
  Interventions: Procedure: distal femoral osteotomies using the PediLoc® Locking Cannulated Blade Plate System
- distal femoral osteotomies using the 90°LCP-PCP
  Interventions: Procedure: distal femoral osteotomies using the 90°LCP-PCP

INTERVENTIONS:
Procedure: distal femoral osteotomies using the PediLoc® Locking Cannulated Blade Plate System — distal femoral osteotomies using the PediLoc® Locking Cannulated Blade Plate System
  Groups: distal femoral osteotomies using the PediLoc® Locking Cannulated Blade Plate System
Procedure: distal femoral osteotomies using the 90°LCP-PCP — distal femoral osteotomies using the 90°LCP-PCP
  Groups: distal femoral osteotomies using the 90°LCP-PCP

SUMMARY:
Background: The PediLoc® Locking Cannulated Blade Plate System, originally designed for proximal femoral osteotomies, has also been used for multidimensional deformity correction of the distal femur. This study describes the surgical technique and retrospectively analyses consolidation rates of distal femoral osteotomies using this system, comparing them to distal femoral osteotomies using the DePuy Synthes® 90°LCP Pediatric Condylar Plate.

Materials and methods: A retrospective review was conducted for patients who underwent distal femoral osteotomy with the PediLoc® Blade Plate (Blade Plate) and the DePuy Synthes® 90°LCP Pediatric Condylar Plate (90°LCP-PCP) at the University Children's Hospital Zurich (2020-2024). Consolidation rates were assessed using Reborn-, Rust-, and modified Rust-scores at 6 weeks, 3 months, and 6 months postoperatively and compared using an unpaired t-test. Geometric planes of osteotomy were analysed, and a stepwise correction technique was described.

ELIGIBILITY:
Inclusion Criteria:

* All Patients that underwent distal femoral osteotomies
* informed consent

Exclusion Criteria:

* intraoperative technical error
* missing data
* missing IC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective study investigated the electronic medical records of patients who underwent distal femoral osteotomy with the Blade Plate system and the 90°LCP-PCP at the University Children's Hospital Zurich between 2020 and 2024.
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Consolidation rates using Reborn-, Rust- and modified Rust-scores on serial X-ray images | 6 weeks, 3 months, 6 months
  Reborn Score: Minimum: 4pts. maximum 16pts., higher scores are better Rust Score ( Radiographic Union Scale for the Tibia ): Minimum: 4pts. maximum 12pts., higher scores are better modified Rust Score ( Radiographic Union Scale for the Tibia ): Minimum: 4pts. maximum 16pts., higher scores are better

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's Hospital Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No